CLINICAL TRIAL: NCT01777074
Title: Measurement of the Changes in Acceptability of Hepatitis B Immunization Among General Practitioners and Open-care Paediatricians
Brief Title: Acceptability of Hepatitis B Vaccination in General Practitioners and Paediatricians
Acronym: PRALINE
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113385
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Hepatitis B
Keywords: Vaccination; Acceptability; Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Generalist physicians Cohort
  Interventions: Other: Data collection
- Paediatricians Cohort
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Questionnaire, Vaccination book

SUMMARY:
The present study is conducted in order to assess the acceptability of Hepatitis B vaccination in French general practitioners and peadiatricians before and after reimbursement of the paediatric vaccine InfanrixHexa. Two data measurement time points are planned, first before reimbursement and after reimbursement.

DETAILED DESCRIPTION:
The aim of the study is to assess the acceptability of Hepatitis B immunization among general practitioners and open-care paediatricians. This is a national, repeated transversal epidemiological study with two data measurement time-points over a period of two years (T1 in 2009, T2 in 2011, two different samples of physicians) in order to assess immunization practices before introduction of the reimbursement of InfanrixHexa®, during the transition period and then during the period following reimbursement of the vaccine. At each collection time-point, two patient age groups will be investigated: 12-15 months and 24-27 months, thus providing measurements before/after reimbursement.

ELIGIBILITY:
Inclusion Criteria:

• Children on the eligibility register complying with the investigator's immunization policy (children followed by the investigator since their birth, whose immunization regimen has been managed by the investigator).

Exclusion Criteria:

* Children on the eligibility register not complying with the investigator's immunization policy.
* Refusal of the patient.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: An eligibility register will be kept throughout the inclusion period by the investigators. All children aged 12 to 15 months and 24 to 27 months, seen by the physician during this period, will be entered on this register General practitioners and open-care paediatricians drawn at random and agreeing to participate in the study.
Sampling Method: Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2009-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of physicians with at least 50% of infants immunized against Hepatitis B. | 4 years

SECONDARY OUTCOMES:
Type of physicians, based on the questionnaire regarding immunization practices and established at each measurement time point. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (368):
- France (368):
  - GSK Investigational Site, Agde
  - GSK Investigational Site, Agen
  - GSK Investigational Site, Aire-sur-la-Lys
  - GSK Investigational Site, Aizenay
  - GSK Investigational Site, Albi
  - GSK Investigational Site, Alès
  - GSK Investigational Site, Alleins
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Ancenis
  - GSK Investigational Site, Andrésy
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Anglet
  - GSK Investigational Site, Annecy
  - GSK Investigational Site, Annecy-le-Vieux
  - GSK Investigational Site, Antony
  - GSK Investigational Site, Argenteuil
  - GSK Investigational Site, Arles
  - GSK Investigational Site, Arnas
  - GSK Investigational Site, Arsac
  - GSK Investigational Site, Asnières-sur-Seine
  - GSK Investigational Site, Aubagne
  - GSK Investigational Site, Aubergenville
  - GSK Investigational Site, Aubervilliers
  - GSK Investigational Site, Aucamville
  - GSK Investigational Site, Auchy-les-Mines
  - GSK Investigational Site, Auriol
  - GSK Investigational Site, Avignon
  - GSK Investigational Site, Bagneux
  - GSK Investigational Site, Bagnols-sur-Cèze
  - GSK Investigational Site, Bar-le-Duc
  - GSK Investigational Site, Barr
  - GSK Investigational Site, Beaulieu-lès-Loches
  - GSK Investigational Site, Beaumont
  - GSK Investigational Site, Beaupréau
  - GSK Investigational Site, Beausoleil
  - GSK Investigational Site, Beauvais
  - GSK Investigational Site, Belfort
  - GSK Investigational Site, Bellegarde
  - GSK Investigational Site, Berre-l'Étang
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Betton
  - GSK Investigational Site, Béthune
  - GSK Investigational Site, Béziers
  - GSK Investigational Site, Biarritz
  - GSK Investigational Site, Bièvres
  - GSK Investigational Site, Biganos
  - GSK Investigational Site, Biscarrosse
  - GSK Investigational Site, Bischheim
  - GSK Investigational Site, Bois-Guillaume
  - GSK Investigational Site, Bollène
  - GSK Investigational Site, Boos
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Bosmie-l'Aiguille
  - GSK Investigational Site, Boulogne-Billancourt
  - GSK Investigational Site, Bourg-en-Bresse
  - GSK Investigational Site, Bousse
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Bron
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Buchy
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Cambrai
  - GSK Investigational Site, Camphin-en-Carembault
  - GSK Investigational Site, Cannes
  - GSK Investigational Site, Carresse-Cassaber
  - GSK Investigational Site, Caveirac
  - GSK Investigational Site, Cergy
  - GSK Investigational Site, Cergy Saint Christophe
  - GSK Investigational Site, Cestas
  - GSK Investigational Site, Chalamont
  - GSK Investigational Site, Challans
  - GSK Investigational Site, Chalon-sur-Saône
  - GSK Investigational Site, Chambly
  - GSK Investigational Site, Champigny-sur-Marne
  - GSK Investigational Site, Chanteloup-les-Vignes
  - GSK Investigational Site, Chantilly
  - GSK Investigational Site, Chartres
  - GSK Investigational Site, Chassieu
  - GSK Investigational Site, Chatou
  - GSK Investigational Site, Châteauneuf-les-Martigues
  - GSK Investigational Site, Châtenois-les-Forges
  - GSK Investigational Site, Cherbourg - Octeville
  - GSK Investigational Site, Clamart
  - GSK Investigational Site, Clapiers
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Clichy
  - GSK Investigational Site, Colmar
  - GSK Investigational Site, Colomars
  - GSK Investigational Site, Colombelles
  - GSK Investigational Site, Combs-la-Ville
  - GSK Investigational Site, Compiègne
  - GSK Investigational Site, Condé-sur-Noireau
  - GSK Investigational Site, Corbeil-Essonnes
  - GSK Investigational Site, Courpière
  - GSK Investigational Site, Creutzwald
  - GSK Investigational Site, Crolles
  - GSK Investigational Site, Cugnaux
  - GSK Investigational Site, Cusset
  - GSK Investigational Site, Darnétal
  - GSK Investigational Site, Deluz
  - GSK Investigational Site, Dessenheim
  - GSK Investigational Site, Digne-les-Bains
  - GSK Investigational Site, Divonne-les-Bains
  - GSK Investigational Site, Domène
  - GSK Investigational Site, Domont
  - GSK Investigational Site, Draguignan
  - GSK Investigational Site, Einvaux
  - GSK Investigational Site, Esquerdes
  - GSK Investigational Site, Essey-lès-Nancy
  - GSK Investigational Site, Estrées-Saint-Denis
  - GSK Investigational Site, Épinal
  - GSK Investigational Site, Équeurdreville-Hainneville
  - GSK Investigational Site, Évreux
  - GSK Investigational Site, Évry
  - GSK Investigational Site, Fenioux
  - GSK Investigational Site, Feurs
  - GSK Investigational Site, Fécamp
  - GSK Investigational Site, Figeac
  - GSK Investigational Site, Fontaine
  - GSK Investigational Site, Fontaine-lès-Dijon
  - GSK Investigational Site, Fontains
  - GSK Investigational Site, Fontenay-sous-Bois
  - GSK Investigational Site, Forges-les-Eaux
  - GSK Investigational Site, Fouesnant
  - GSK Investigational Site, Foussais-Payré
  - GSK Investigational Site, Francheville
  - GSK Investigational Site, Fumel
  - GSK Investigational Site, Gamarde-les-Bains
  - GSK Investigational Site, Gémozac
  - GSK Investigational Site, Gondecourt
  - GSK Investigational Site, Gonneville-la-Mallet
  - GSK Investigational Site, Gouvieux
  - GSK Investigational Site, Gouy-sous-Bellonne
  - GSK Investigational Site, Gouzeaucourt
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Gréoux-les-Bains
  - GSK Investigational Site, Grigny
  - GSK Investigational Site, Guénange
  - GSK Investigational Site, Haguenau
  - GSK Investigational Site, Hatten
  - GSK Investigational Site, Hesdin
  - GSK Investigational Site, Houilles
  - GSK Investigational Site, Houplin-Ancoisne
  - GSK Investigational Site, Hyères
  - GSK Investigational Site, Hœnheim
  - GSK Investigational Site, Illkirch-Graffenstaden
  - GSK Investigational Site, Istres
  - GSK Investigational Site, Jarny
  - GSK Investigational Site, Joué-lès-Tours
  - GSK Investigational Site, L'Aigle
  - GSK Investigational Site, L'Huisserie
  - GSK Investigational Site, La Chapelle-sur-Erdre
  - GSK Investigational Site, La Couronne
  - GSK Investigational Site, La Crèche
  - GSK Investigational Site, La Garenne-Colombes
  - GSK Investigational Site, La Madeleine
  - GSK Investigational Site, La Mézière
  - GSK Investigational Site, La Motte-Servolex
  - GSK Investigational Site, La Source Orleans
  - GSK Investigational Site, La Talaudière
  - GSK Investigational Site, La Voulte-sur-Rhône
  - GSK Investigational Site, Lamarche-sur-Saône
  - GSK Investigational Site, Lambersart
  - GSK Investigational Site, Landivisiau
  - GSK Investigational Site, Lanester
  - GSK Investigational Site, Langon
  - GSK Investigational Site, Laval
  - GSK Investigational Site, Le Barp
  - GSK Investigational Site, Le Bouscat
  - GSK Investigational Site, Le Cannet
  - GSK Investigational Site, Le Chesnay
  - GSK Investigational Site, Le Creusot
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Le Lavandou
  - GSK Investigational Site, Le Palais-sur-Vienne
  - GSK Investigational Site, Le Passage D' Agen
  - GSK Investigational Site, Le Rheu
  - GSK Investigational Site, Les Sables-d'Olonne
  - GSK Investigational Site, Les Ulis
  - GSK Investigational Site, Lesquin
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Limas
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Lingolsheim
  - GSK Investigational Site, Lisieux
  - GSK Investigational Site, Lognes
  - GSK Investigational Site, Lomme
  - GSK Investigational Site, Loos-en-Gohelle
  - GSK Investigational Site, Lorient
  - GSK Investigational Site, Luzinay
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Malakoff
  - GSK Investigational Site, Mantes-la-Ville
  - GSK Investigational Site, Marchenoir
  - GSK Investigational Site, Marcq-en-Barœul
  - GSK Investigational Site, Marguerittes
  - GSK Investigational Site, Marmande
  - GSK Investigational Site, Marnay
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Martigues
  - GSK Investigational Site, Martin-Église
  - GSK Investigational Site, Martinsart
  - GSK Investigational Site, Mauze Sur Mignon
  - GSK Investigational Site, Meaux
  - GSK Investigational Site, Merkwiller-Pechelbronn
  - GSK Investigational Site, Metz
  - GSK Investigational Site, Meudon
  - GSK Investigational Site, Meylan
  - GSK Investigational Site, Meyssac
  - GSK Investigational Site, Mérignac
  - GSK Investigational Site, Méry-sur-Oise
  - GSK Investigational Site, Mirecourt
  - GSK Investigational Site, Moivrons
  - GSK Investigational Site, Molsheim
  - GSK Investigational Site, Mondeville
  - GSK Investigational Site, Mons-en-Barœul
  - GSK Investigational Site, Montauban
  - GSK Investigational Site, Monteux
  - GSK Investigational Site, Montélimar
  - GSK Investigational Site, Montfermeil
  - GSK Investigational Site, Montgeron
  - GSK Investigational Site, Montigny-le-Bretonneux
  - GSK Investigational Site, Montigny-lès-Metz
  - GSK Investigational Site, Montoire-sur-le-Loir
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Montreuil
  - GSK Investigational Site, Morlaàs
  - GSK Investigational Site, Morlaix
  - GSK Investigational Site, Mornas
  - GSK Investigational Site, Mouans-Sartoux
  - GSK Investigational Site, Moutiers Tarentaise
  - GSK Investigational Site, Moyeuvre-Grande
  - GSK Investigational Site, Mur-de-Sologne
  - GSK Investigational Site, Nanterre
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nemours
  - GSK Investigational Site, Neuville-sur-Saône
  - GSK Investigational Site, Niort
  - GSK Investigational Site, Nogent-sur-Marne
  - GSK Investigational Site, Noisy-le-Roi
  - GSK Investigational Site, Noyon
  - GSK Investigational Site, Obernai
  - GSK Investigational Site, Oloron-Sainte-Marie
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Orthez
  - GSK Investigational Site, Oucques
  - GSK Investigational Site, Ouistreham
  - GSK Investigational Site, Oust
  - GSK Investigational Site, Ozoir-la-Ferrière
  - GSK Investigational Site, Palaiseau
  - GSK Investigational Site, Pamiers
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pau
  - GSK Investigational Site, Pertuis
  - GSK Investigational Site, Pierrefitte-sur-Sauldre
  - GSK Investigational Site, Plouguernével
  - GSK Investigational Site, Pont Ste Maxence
  - GSK Investigational Site, Pont-à-Mousson
  - GSK Investigational Site, Pont-l'Abbé-d'Arnoult
  - GSK Investigational Site, Pontarlier
  - GSK Investigational Site, Pornic
  - GSK Investigational Site, Port-sur-Saône
  - GSK Investigational Site, Provins
  - GSK Investigational Site, Publier
  - GSK Investigational Site, Puteaux
  - GSK Investigational Site, Quévreville-la-Poterie
  - GSK Investigational Site, Râches
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Rezé
  - GSK Investigational Site, Rillieux-la-Pape
  - GSK Investigational Site, Riom
  - GSK Investigational Site, Rivery
  - GSK Investigational Site, Roanne
  - GSK Investigational Site, Roche-la-Molière
  - GSK Investigational Site, Rodez
  - GSK Investigational Site, Romainville
  - GSK Investigational Site, Romans-sur-Isère
  - GSK Investigational Site, Romillé
  - GSK Investigational Site, Ronchin
  - GSK Investigational Site, Rosières-en-Santerre
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Royan
  - GSK Investigational Site, Ruy
  - GSK Investigational Site, Sahurs
  - GSK Investigational Site, Saint-Astier
  - GSK Investigational Site, Saint-Aubin
  - GSK Investigational Site, Saint-Aubin-sur-Scie
  - GSK Investigational Site, Saint-Brevin-les-Pins
  - GSK Investigational Site, Saint-Brieuc
  - GSK Investigational Site, Saint-Chamond
  - GSK Investigational Site, Saint-Chéron
  - GSK Investigational Site, Saint-Cloud
  - GSK Investigational Site, Saint-Cyr-au-Mont-d'Or
  - GSK Investigational Site, Saint-Denis
  - GSK Investigational Site, Saint-Etienne
  - GSK Investigational Site, Saint-Étienne-de-Montluc
  - GSK Investigational Site, Saint-Flour
  - GSK Investigational Site, Saint-Genis-Laval
  - GSK Investigational Site, Saint-Germain-lès-Arpajon
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Saint-Ismier
  - GSK Investigational Site, Saint-Jean-de-la-Ruelle
  - GSK Investigational Site, Saint-Leu-la-Forêt
  - GSK Investigational Site, Saint-Louis
  - GSK Investigational Site, Saint-Loup-sur-Semouse
  - GSK Investigational Site, Saint-Nazaire
  - GSK Investigational Site, Saint-Pierre-d'Irube
  - GSK Investigational Site, Saint-Pol-sur-Mer
  - GSK Investigational Site, Saint-Priest
  - GSK Investigational Site, Saint-Rémy-de-Provence
  - GSK Investigational Site, Saint-Tropez
  - GSK Investigational Site, Saintes
  - GSK Investigational Site, Sanary-sur-Mer
  - GSK Investigational Site, Segonzac
  - GSK Investigational Site, Segré
  - GSK Investigational Site, Sens
  - GSK Investigational Site, Septèmes-les-Vallons
  - GSK Investigational Site, Serres
  - GSK Investigational Site, Sélestat
  - GSK Investigational Site, Sillery
  - GSK Investigational Site, Soissons
  - GSK Investigational Site, Sorgues
  - GSK Investigational Site, St-Malo
  - GSK Investigational Site, St.-Jean
  - GSK Investigational Site, Ste Foy La Grande
  - GSK Investigational Site, Ste Maxime
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Sucy-en-Brie
  - GSK Investigational Site, Suresnes
  - GSK Investigational Site, Talence
  - GSK Investigational Site, Tarascon
  - GSK Investigational Site, Thiais
  - GSK Investigational Site, Thonon-les-Bains
  - GSK Investigational Site, Thun-Saint-Amand
  - GSK Investigational Site, Toul
  - GSK Investigational Site, Toulon
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Trie-Château
  - GSK Investigational Site, Troyes
  - GSK Investigational Site, Vabres-l'Abbaye
  - GSK Investigational Site, Val-de-Vesle
  - GSK Investigational Site, Valence
  - GSK Investigational Site, Vallauris
  - GSK Investigational Site, Vandœuvre-lès-Nancy
  - GSK Investigational Site, Vannes
  - GSK Investigational Site, Vaugneray
  - GSK Investigational Site, Vaulx-en-Velin
  - GSK Investigational Site, Vauréal
  - GSK Investigational Site, Vaux-le-Pénil
  - GSK Investigational Site, Vendargues
  - GSK Investigational Site, Vernouillet
  - GSK Investigational Site, Versailles
  - GSK Investigational Site, Vertou
  - GSK Investigational Site, Villars-les-Dombes
  - GSK Investigational Site, Villeblevin
  - GSK Investigational Site, Villeneuve-d'Ascq
  - GSK Investigational Site, Villeurbanne
  - GSK Investigational Site, Villiers-sur-Marne
  - GSK Investigational Site, Vincennes
  - GSK Investigational Site, Viry-Châtillon
  - GSK Investigational Site, Vitrolles
  - GSK Investigational Site, Vitry-sur-Seine
  - GSK Investigational Site, Voreppe
  - GSK Investigational Site, Wattignies
  - GSK Investigational Site, Yerres
  - GSK Investigational Site, Zillisheim